CLINICAL TRIAL: NCT02498002
Title: Impacts of Intermittent Fasting in Adults on Energy Balance, Body Composition, Postprandial Hormone Profiles and Gene Expression in Adipose Tissue
Brief Title: Impacts of Intermittent Fasting on Energy Balance and Associated Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Betts, Professor of Metabolic Physiology, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMF-02
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Diet; Fasting; Intermittent Fasting; Alternate-day Fasting; Physical Activity; Glucose; Insulin; Appetite
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Fasting; Intermittent Fasting; Motor Activity; Insulin Resistance | interventions — Lidocaine; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daily Calorie Restriction (DCR) (Active Comparator): During the intervention phase, participants randomised to this treatment condition will be asked to reduce their normal energy intake by 25% on a daily basis.
  Interventions: Device: Physical Activity Monitoring (Actiheart); Other: Energy Intake Monitoring; Other: Body Weight Monitoring; Procedure: Intravenous Cannulation; Procedure: Adipose Tissue Biopsy; Drug: Lidocaine Hydrochloride; Other: Post-Prandial Meal Tests; Radiation: DEXA Scan; Other: Actiheart Calibration; Other: Daily Calorie Restriction
- Fasting with Weight Loss (IMF-WL) (Experimental): During the intervention phase, participants randomised to this treatment condition will be asked to alternate between 24 hour cycles of feeding (consume 150% of normal energy intake) and fasting (no energy intake).
  Interventions: Device: Physical Activity Monitoring (Actiheart); Other: Energy Intake Monitoring; Other: Body Weight Monitoring; Procedure: Intravenous Cannulation; Procedure: Adipose Tissue Biopsy; Drug: Lidocaine Hydrochloride; Other: Post-Prandial Meal Tests; Radiation: DEXA Scan; Other: Actiheart Calibration; Other: Intermittent Fasting with Weight Loss
- Fasting without Weight Loss (IMF-WS) (Experimental): During the intervention phase, participants randomised to this treatment condition will be asked to alternate between 24 hour cycles of feeding (consume 200% of normal energy intake) and fasting (no energy intake).
  Interventions: Device: Physical Activity Monitoring (Actiheart); Other: Energy Intake Monitoring; Other: Body Weight Monitoring; Procedure: Intravenous Cannulation; Procedure: Adipose Tissue Biopsy; Drug: Lidocaine Hydrochloride; Other: Post-Prandial Meal Tests; Radiation: DEXA Scan; Other: Actiheart Calibration; Other: Intermittent Fasting without Weight Loss

INTERVENTIONS:
Device: Physical Activity Monitoring (Actiheart) — Monitor physical activity using an Actiheart monitor during the required periods.
Other: Energy Intake Monitoring — Monitor energy intake by weighing and recording all foods/drinks consumed during the required periods.
Other: Body Weight Monitoring — Monitor body weight during monitoring phase to ensure stability despite other monitoring activities.
Procedure: Intravenous Cannulation — Fitting of an intravenous cannula to a vein on the forearm for blood sampling during laboratory protocols.
Procedure: Adipose Tissue Biopsy — This is an optional feature which if included involves the removal of a 0.5 gram sample of adipose tissue from just below the skin using a needle.
Drug: Lidocaine Hydrochloride — The anaesthetic that will be used to numb the site of the adipose tissue biopsy in the event it is included.
Other: Post-Prandial Meal Tests — Consume two successive meals with regular blood samples throughout the ensuing hours (2-3 hours each).
Radiation: DEXA Scan — Undergo a dual energy x-ray absorptiometry scan to examine body composition.
Other: Actiheart Calibration — Submaximal treadmill test to calibrate monitoring equipment.
Other: Daily Calorie Restriction — Reduce energy intake by 25% on a daily basis.
  Arms: Daily Calorie Restriction (DCR)
Other: Intermittent Fasting with Weight Loss — Alternate between 24 hour cycles of fasting and feeding with 150% of normal intake when feeding.
  Arms: Fasting with Weight Loss (IMF-WL)
Other: Intermittent Fasting without Weight Loss — Alternate between 24 hour cycles of fasting and feeding with 200% of normal intake when feeding.
  Arms: Fasting without Weight Loss (IMF-WS)

SUMMARY:
Obesity is a global concern with links to conditions such as diabetes. Historically, these conditions have been managed by reducing energy intake on a daily basis, which is often hampered by low adherence rates and compensatory reductions in physical activity. Intermittent fasting (IMF) has become popular as an alternative method of weight loss, where periods of normal eating are punctuated by days of fasting. However, despite its popularity, IMF is scarcely examined within the literature.

This study will examine the impact of IMF on energy balance and the associated health outcomes relating to conditions such as diabetes. To achieve this, 36 lean adults and 36 overweight/obese adults will be recruited, excluding those with conditions which may be adversely affected by fasting. Once enrolled, participants will complete a one month control phase, incorporating 12 days of diet and activity monitoring, to ensure their weight is stable before moving in to the intervention phase.

The intervention phase will begin with a lab protocol designed to examine body composition, resting metabolic rate and metabolic responses to two successive meals. Once completed, participants will be randomised to one of three diets which are listed below. Comparing the changes seen with diets 1 and 2 will provide the first direct comparison of IMF against more conventional strategies, while diet 3 will allow us to ascertain the role of weight loss in mediating any effects of IMF.

1. Daily calorie restriction - Reduce energy intake by 25% on a daily basis
2. IMF with weight loss - Alternate between 24 hour cycles of fasting and feeding with 150% of normal intake when feeding
3. IMF without weight loss - Alternate between 24 hour cycles of fasting and feeding with 200% of normal intake when feeding

All three diets will last for 20 consecutive days, with transitions between each 24 hour diet cycle occurring at 15:00 each day to allow at least one main meal per day. When fasting, participants will only be permitted water and black tea/coffee to eliminate energy intake. Once again physical activity and diet will be monitored for 12 days during the intervention to examine changes in energy expenditure and ensure compliance.

Having completed all 20 diet cycles participants will return to the laboratory to repeat the protocol described earlier. Comparing these results against the values seen before the intervention will then allow the effects of IMF to be identified and compared.

DETAILED DESCRIPTION:
Recruitment

Local advertising in the form of posters will distributed throughout the research institution, nearby organisations and the city of Bath. The posters will encourage interested persons to contact the chief investigator to receive more information on what the study will involve. The research team will be looking to recruit 72 (36 lean, 36 overweight/obese) individuals who satisfy the entry criteria (discussed later).

Enrolment

Potential volunteers will use the contact details provided in advertising materials to express their interest to the research team who will then provide them with a copy of the participant information sheet to read through at their convenience. Those interested in participating will then be invited to a pre-enrolment consultation where they will be given the opportunity to ask any questions they may have about the study before being screened for the inclusion and exclusion criteria. This will involve measurements of weight and height, as well as the completion of an entry criteria questionnaire, the Eating Disorder Examination Questionnaire and the Physical Activity Readiness Questionnaire. Providing they satisfy the relevant criteria they will be talked through the study and before being asked to complete an informed consent form. As part of this, the procedure for an adipose tissue biopsy will be discussed with the participant and they will be asked to decide whether or not they would like to include this as it is an optional test.

Baseline Lab Protocol (LAB 1)

Having formally enrolled in the study, participants will be invited to begin their involvement in the study with a 60 minute visit to the University of Bath following a 12 hour fast. During this visit, the researcher will obtain a urine sample to check hydration levels using an Osmometer, before taking measurements of height, weight and waist circumference. A fasting blood sample will also be obtained using venepuncture to measure resting levels of key hormones and metabolites. To conclude this visit participants will be asked to perform a submaximal exercise test to calibrate the 'Actiheart' monitor being used throughout the study to measure physical activity energy expenditure. For this, participants will be asked to remain on a treadmill as the intensity increases over the following four stages:

* Stage 1 - level walking at 3.2 km/h
* Stage 2 - brisk walking at 5.2 km/h
* Stage 3 - brisk walking at 5.8 km/h with a steep gradient of +10.2%
* Stage 4 - level running at 12.5 km/h

Stage 4 will only be included for those who are formal exercisers, as non-exercisers are unlikely to be doing this kind of activity in their normal routine rendering a calibration at this intensity unnecessary. Formal exercisers will be identified using the entry criteria questionnaire. In addition, the treadmill protocol will be stopped earlier if the participant asks to stop or if their heart rate exceeds 85% of their age-predicted maximum.

Monitoring Phase

Before leaving the lab, participants will be provided with an Actiheart monitor, a small device applied to the chest which measures physical activity by recording heart rate and movement every minute. They will also be provided with a set of kitchen scales and a log book to create a weighed record of their food and fluid intake and a set of body weight scales to track their weight and help keep it stable.

During the four week monitoring phase, participants will be asked to complete four 3-day monitoring periods, each comprising two weekdays and one weekend day whilst they continue in their normal dietary and exercise habits. The researchers will arrange the collection and delivery of monitoring equipment where necessary. The purpose of this is firstly to ensure weight stability to minimise any confounding influences, secondly to provide accurate baseline values for key variables such as physical activity, and finally to ensure the dietary records provided are a valid reflection of habitual intake.

Provided the data obtained in the control phase satisfies the relevant reliability criteria, participants will be invited to return to the physiology lab at least four weeks after their first visit. In preparation for this, participants will be asked to avoid strenuous exercise, alcohol and caffeine, before fasting overnight until they arrive at the lab the following morning.

Pre-Intervention Lab Protocol (LAB 2)

Before beginning their intervention participants will be asked to attend a pre-intervention lab protocol, as outlined below. Female participants will be asked to schedule this so that it coincides with the follicular phase of their menstrual cycle (3-10 days after the onset of menses) as this is when their hormone profiles are at their most stable.

On the day of their visit participants will be asked to consume one pint of water at 06:30 before preparing themselves to arrive at the lab by 07:30, wearing light clothes (i.e. shorts, t-shirt) with no metal components or jewellery. They will then need to provide a small urine sample to check hydration levels before measurements of height, weight and waist circumference are taken (NOTE: If weight varies by more than 1.0 kilograms compared to their baseline measurement they may be asked to repeat the monitoring phase).

At 07:45 participants will be asked to lie in a semi-recumbent position and rest for 30 minutes. This is in preparation for the measurement of resting metabolic rate and substrate oxidation which will be completed at 08:15 over three 5-minute periods using indirect calorimetry while the participant remains rested. Following this an intravenous cannula will be fitted to the antecubital vein at the elbow for blood sampling throughout the visit. At this point a 12 ml fasting blood sample will also be drawn to measure resting levels of key metabolites (e.g. glucose, insulin, cholesterol, leptin, ghrelin, etc.).

At 08:45, participants who have elected to include the adipose tissue biopsy will undergo this procedure. If included, an area on the side of the abdomen just above the waistband will be sterilised and injected with an anaesthetic (Lidocaine Hydrochloride) to numb the area. Using a larger needle a 0.5 gram sample of adipose tissue will then be taken from just below the skin. There will some bruising, but if left to heal there should be no scarring. Those who choose not to include this biopsy will simply continue resting.

At 09:00 participants will be asked to complete visual analogue scales (VAS) which will provide subjective measures of appetite, fullness and desire to eat. Immediately after this, participants will be provided with a test breakfast of instant porridge made with whole milk and sugar which they will need to consume within 10 minutes. Key measures will then be taken at the following intervals:

* 12 ml blood sample - 15, 30, 45, 60, 90, 120, 180
* Visual analogue scales - 30, 60, 90, 120, 150, 180
* Metabolic rate (indirect calorimetry) - 60. 120, 180

(Note: total urine output will also be quantified throughout the postprandial period to adjust substrate oxidation values for protein oxidation)

At 12:05 participants will be asked to place the hand of their cannulated arm in a padded Perspex box which will be heated to 55 degrees. This is to allow the venous blood to be arterialised which will provide a better indication of whole body glucose metabolism in the test which follows. At 12:15 a 7 ml blood sample will be drawn after which the participant will be asked to consume a milkshake which provides 33% of their energy requirements. Blood samples (7 ml) will then be drawn every 15 minutes for the ensuing two hours to test for the presence of a second meal effect. At 14:15 the final blood sample for this visit will be drawn and the cannula will be removed.

To conclude the pre-intervention protocol participants will be taken to a separate lab for a dual-energy x-ray absorptiometry (DEXA) scan. This is a specialized form of whole-body scan which measures how a person's weight is distributed between fat and muscle tissue. It takes approximately eight minutes and requires the participant to lie still throughout. It does administer a small dose of ionizing radiation, but this is equivalent to 7 microSieverts which is accompanied by a risk of detrimental radiation effects in the region of 1 in 10 million. The application of this method has been approved in this study by an independent medical physics expert and a clinical radiation expert.

Intervention Phase

Before exiting the lab participants will be randomised to one of three treatment conditions outlined below. All three diet groups will last for 20 days in total, with transitions between each 24 hour cycle occurring at 15:00 each day, the idea being that it will allow them to consume at least one main meal per day in all cases. For the intermittent fasting groups (IMF), please note that during fasted cycles participants will be asked to only consume water and black tea/coffee with no milk or sugar. During feeding cycles, and throughout the daily calorie restriction diet, participants will be asked to recreate their control phase diet record with appropriately modified quantities to give 75%, 150% or 200% of their normal calorie intake in accordance with the group they are assigned to. Where recreation is not possible, participants will be asked to note the item that has been removed and/or the item that was added in a new diet record that will be provided before they leave the lab. Physical activity will also be monitored for the first and last week of the intervention using an Actiheart monitor to examine behavioural adaptations to the diets.

1. Daily calorie restriction - Reduce energy intake by 25% on a daily basis
2. IMF with weight loss - Alternate between 24 hour cycles of fasting and feeding with 150% of normal intake when feeding
3. IMF without weight loss - Alternate between 24 hour cycles of fasting and feeding with 200% of normal intake when feeding

At 15:00 on the day of their initial lab visit, male participants will begin their assigned diet, although this can be postponed by up to one week if necessary. Female participants will be asked to delay this by six days in all cases in order to ensure their post-intervention lab visit falls within the same phase of their menstrual cycle to minimise the impact of monthly hormonal fluctuations.

Post-Intervention Lab Protocol (LAB 3)

Following the completion of 20 consecutive 24 hour dietary cycles, participants will return to their normal diet for one day (prescribed) whilst avoiding strenuous exercise, smoking, alcohol and caffeine, before fasting until they arrive at the lab the following morning for their post-intervention lab visit. Having consumed a pint of water at 06:30 and arrived at 07:30 in light clothing, participants will undergo the same lab protocol described earlier for their pre-intervention visit. However, instead of being randomised to a diet group they will be asked to complete a feedback questionnaire on their experience of the study.

Follow-up

Four weeks after their post-intervention lab visit participants will be invited to a feedback session to discuss all available results. The results from the meal test and the study as a whole will follow at a later date due to logistics and cost-effectiveness. Where convenient participants will also be asked to include a weight measurement to provide an indication of weight loss sustainability.

Aim

Once datasets are obtained for all 72 participants, the daily calorie restriction group will be compared against the IMF with weight loss group. This will permit the comparison of the effects of an IMF diet against the effects of a more conventional approach when matched for energy deficit. The final group, IMF without weight loss, will then highlight the relative contributions of weight loss and fasting-dependent mechanisms in producing any observed effects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 20.5 kg/m2 or greater
* Stable body weight for preceding three months (<3 kg increase or decrease)
* Able and willing to safely comply with study procedures
* Be able to attend the laboratory and willing to participate in necessary protocols
* Be willing to undertake the durations of fasting required by the study
* Have the capacity and willingness to provide informed consent (oral and written)

Exclusion Criteria:

* Have a body weight greater than 120 kg
* Will be undertaking any other fasting practices during their participation in the study (can enrol once stable weight returns after fasting is completed)
* Currently engaged in or planning to engage in another weight management programme (e.g. weight watchers) or exercise programme (e.g. hypertrophy training or marathon training) during the study
* Have previously suffered or are suffering from an eating disorder as assessed using the Eating Disorder Examination Questionnaire, Version 6.0 (Fairburn & Beglin, 2008)
* Have been diagnosed with either type 1 or type 2 diabetes
* Undertaking any form of medical treatment which may interfere with study variables (e.g. chemotherapy, liposuction, taking metformin, statins/other lipid-lowering medications)
* Are peri-menopausal or menopausal (absence of menses for 3-24 months)
* Pregnant, recently pregnant (within last 6 months), planning to become pregnant (within next six months), or currently breastfeeding.
* Have donated more than 500 ml of blood in the last three months before the initial laboratory visit
* Lack of metal capacity or language skills to independently understand/follow the study protocol
* Physical disability which impacts study variables or ability to independently follow study protocol (e.g. paralysis)
* Cannot consume test meals due to intolerances (i.e. lactose)
* Report medical contraindications on the 'Physical Activity Readiness Questionnaire' and are unable to obtain medical approval for the treadmill test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage | Pre - Post (3 weeks)
  Comparison of body fat percentage (measured by dual-energy x-ray absorptiometry) from pre-intervention time-point to post-intervention time-point.
Lean Body Mass | Pre - Post (3 weeks)
  Comparison of lean body mass (measured by dual-energy x-ray absorptiometry) from pre-intervention time-point to post-intervention time-point.
Fasting Plasma Glucose Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of glucose concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting Plasma Insulin Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of insulin concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting Plasma Triglyceride Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of triglyceride concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting Total Cholesterol Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of total cholesterol concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting LDL Cholesterol Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of LDL cholesterol concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting HDL Cholesterol Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of HDL cholesterol concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting Leptin Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of leptin concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting Adiponectin Concentration | Baseline - Pre - Post (7 weeks)
  Comparison of adiponectin concentration in the blood plasma at rest across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Fasting Resting Metabolic Rate | Baseline - Pre - Post (7 weeks)
  Comparison of resting metabolic rate (measured by indirect calorimetry) across all three measurement points to ensure stability in the monitoring phase and examine change during the intervention phase.
Post-Prandial Glucose AUC | Pre - Post (3 weeks)
  Comparison of the area under the plasma glucose curve seen during the 180 minute post-prandial period following a test meal conducted before and after the intervention phase.
Post-Prandial Insulin AUC | Pre - Post (3 weeks)
  Comparison of the area under the plasma insulin curve seen during the 180 minute post-prandial period following a test meal conducted before and after the intervention phase.
Post-Prandial Ghrelin AUC | Pre - Post (3 weeks)
  Comparison of the area under the plasma ghrelin curve seen during the 180 minute post-prandial period following a test meal conducted before and after the intervention phase.
Post-Prandial Peptide-YY AUC | Pre - Post (3 weeks)
  Comparison of the area under the plasma peptide-YY curve seen during the 180 minute post-prandial period following a test meal conducted before and after the intervention phase.
Physical Activity Energy Expenditure | Monitoring - Intervention (7 weeks)
  Comparison of the mean physical activity energy expenditure values recorded using the Actiheart monitor during the monitoring and intervention phase to see the impact of the three treatments on physically active behaviours.
Physical Activity Intensity | Monitoring - Intervention (7 weeks)
  Comparison of the mean physical activity intensity values recorded using the Actiheart monitor during the monitoring and intervention phase to see the impact of the three treatments on physically active behaviours.
CLOCK Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
NPAS2 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PER1 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
CRY1 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
LEP Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
ADIPO-Q Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
IL-6 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
TNF Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
LPL Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
FABP4 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PPARG Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PPARGC1A Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
SREBP1C Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
FSP27 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PRKAA1 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
ANGPTL4 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
HSL Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
ATGL Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PNPLA3 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
CIDE-A Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
GLUT-4 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
AKT2 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PDK4 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
SIRT1 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
SIRT3 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
UCP2 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
IGF1R Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
IRS1 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
IRS2 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
PIK3R1 Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
ChREBP Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
ACACA Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
FASN Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)
ACADM Gene Expression in Subcutaneous Adipose Tissue | Pre - Post (3 weeks)

SECONDARY OUTCOMES:
Fasting Carbohydrate Oxidation | Pre - Post (3 weeks)
  Comparison of carbohydrate oxidation rate measured by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.
Fasting Lipid Oxidation | Pre - Post (3 weeks)
  Comparison of lipid oxidation rate measured by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.
Fasting Protein Oxidation | Pre - Post (3 weeks)
  Comparison of protein oxidation rate measured by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.
Post-Prandial Resting Metabolic Rate | Pre-intervention 60, 120 and 180 minutes after meal - post-intervention 60, 120 and 180 minutes after meal (3 weeks)
  Comparison of post-prandial metabolic rate measured 60, 120 and 180 minutes after a test meal by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.
Post-Prandial Carbohydrate Oxidation | Pre-intervention 60, 120 and 180 minutes after meal - post-intervention 60, 120 and 180 minutes after meal (3 weeks)
  Comparison of post-prandial carbohydrate oxidation rate measured 60, 120 and 180 minutes after a test meal by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.
Post-Prandial Lipid Oxidation | Pre-intervention 60, 120 and 180 minutes after meal - post-intervention 60, 120 and 180 minutes after meal (3 weeks)
  Comparison of post-prandial lipid oxidation rate measured 60, 120 and 180 minutes after a test meal by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.
Post-Prandial Protein Oxidation | Pre-intervention 60, 120 and 180 minutes after meal - post-intervention 60, 120 and 180 minutes after meal (3 weeks)
  Comparison of post-prandial protein oxidation rate measured 60, 120 and 180 minutes after a test meal by indirect calorimetry before and after the intervention phase to examine the effect of the three treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: James A Betts, BSc., Ph.D, Principal Investigator — Fellow of the American College of Sports Medicine
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

REFERENCES:
- [Derived] Templeman I, Thompson D, Gonzalez J, Walhin JP, Reeves S, Rogers PJ, Brunstrom JM, Karagounis LG, Tsintzas K, Betts JA. Intermittent fasting, energy balance and associated health outcomes in adults: study protocol for a randomised controlled trial. Trials. 2018 Feb 2;19(1):86. doi: 10.1186/s13063-018-2451-8. PMID 29394908